CLINICAL TRIAL: NCT02791347
Title: Nutrition Intervention Among Stem Cell Recipients: a Randomized Controlled Trial Post Hospital Discharge
Brief Title: Nutrition Intervention Among Stem Cell Recipients: Post Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Aix Marseille Université (Other)
Responsible Party: Principal Investigator, Jean El Sheikh, Assistant Professor of Hematology Oncology- Department of Internal Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IM.J-EC.01
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Hematopoietic Stem Cell Transplantation; Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Upon discharge from the medical center, patients would be advised on a qualitative, neutropenic diet. Participants' quality of life, physical activity level, functional and nutritional status would be assessed at days +30, +60 and +100 post transplantation.
  These participants will not receive nutritional counseling by the dietitian as outpatients except if referred by the medical team.
- Nutrition Intervention Group (Experimental): Upon discharge from the medical center, NIG patients will receive tailored nutrition counseling with the provision of patient education material and oral nutritional supplements if needed. Patients will be advised on a diet high in energy and proteins and tailored to their medical condition in the hospital before discharge.
  Patients will be followed up at days +30, +60 and +100 post transplantation. Compliance will be measured at each visit by comparing patients caloric and protein needs to their actual protein and energy intake. Compliance will be reinforced to meet patients' goals using nutritional tips, oral supplementation, and artificial nutrition use.
  Interventions: Other: Nutrition Intervention

INTERVENTIONS:
Other: Nutrition Intervention
  Arms: Nutrition Intervention Group

SUMMARY:
Chemotherapy conditioning, preceding Stem Cell Transplantation (SCT), has been associated with severe gastrointestinal toxicity, commonly compromising patients' food intake, nutritional status and functioning level. Malnutrition has been associated with worse functional status, reduced survival, increased rate of infections, complications, hospitalizations, and therapy toxicity in oncology patients.

To date, there is no Randomized Controlled Trials (RCT) assessing the impact of a nutrition intervention on SCT patients who remain at risk of malnutrition even 100 days post SCT. The proposed study is a single center, prospective, RCT with a parallel design that aims to assess the impact of a nutrition intervention on the nutritional and functional statuses of SCT recipients 100 days post SCT.

DETAILED DESCRIPTION:
This study is a single center RCT with a parallel design. It aims to improve the SCT recipients' nutritional status and QoL and reduce the associated morbidities. Results of the study can guide the recommendations for the medical and nutritional outpatient assessment post SCT.

During the pre-SCT workup, patients will be invited to participate in the study. Around discharge from the hospital, recruited patients will be randomized to a control or an intervention group based on permuted block random sampling. Patients in the Nutrition Intervention group (NIG) will receive a tailored diet plan from the dietitian as well as regular outpatient follow-ups measuring and reinforcing compliance. Patients in the Control Group (CG) will receive usual care; they will only be assessed in the nutrition clinics upon referral by the medical team. The body composition, Quality of Life (QoL), Physical Activity (PA) level, nutrient intake, functional status and nutritional status of both groups will be evaluated at regular intervals during the hospital stay and post discharge through the Patient Generated Subjective Global Assessment (PGSGA), Body Impedance Analysis (BIA), handgrip strength, Functional Assessment of Cancer Therapy -Bone Marrow Transplantation (FACT-BMT), PA questionnaire and Karnofsky scale. Moreover, patients' food intake will be analyzed for its micronutrient and macronutrient content to assess the changes in nutrient analysis in the peri-transplantation phase. When applicable, BIA and Computed Tomography (CT) tests will be compared for their agreements.

Considering a power of 80%, an attrition rate of 30% and a difference of 40% between the NIG and CG groups, 52 patients need to be recruited in the study. Analysis will be done based on 'intention to treat' and 'per protocol' analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to the adult BMT service at AUBMC
* Allogeneic or autologous SCT
* Malignant or non-malignant indication for SCT

Exclusion Criteria:

* Patients who pass away before day +100
* Patients who miss 2 assessment points

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a PGSGA score ≥4 | 100 days post transplantation

SECONDARY OUTCOMES:
Handgrip strength | 100 days post transplantation
Lean Body Mass Changes | 100 days post transplantation
Re-hospitalization Rate | 100 days post transplantation
Quality of life (QoL) [ Time Frame: 100 days post transplantation ] | 100 days post transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon